CLINICAL TRIAL: NCT00950976
Title: Clinical Trial of Enteral Citrulline in Volunteers With Surgical Repair of Ventral Hernias
Brief Title: Dose-response Enteral Citrulline for Normal Healthy Volunteers and Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ACSC-CIT-04-06-US
Record Dates: First submitted 2009-07-10; First posted 2009-08-03 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Nutritional Deficiency
MeSH Terms: conditions — Malnutrition | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citrulline (Experimental)
  Interventions: Other: citrulline
- lemonade (Placebo Comparator): Equal volume and flavor to citrulline.
  Interventions: Other: Lemonade

INTERVENTIONS:
Other: citrulline — TID for 5 days
  Arms: Citrulline
Other: Lemonade — TID for 5 days
  Arms: lemonade

SUMMARY:
To determine the level of citrulline to produce a given amount of arginine in healthy volunteers and surgical patients. Arginine-related amino acids are expected to increase as a result of increased substrate provided by citrulline.

ELIGIBILITY:
Inclusion Criteria:

* adults, male & female, non-pregnant
* BMI 18.5-29.9

Exclusion Criteria:

* cancer
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-03; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Plasma amino acid levels | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Juan B. Ochoa, MD Prof., Principal Investigator — Associate Professor of Surgery and Critical Care, University of Pittsburgh Physicians
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States